CLINICAL TRIAL: NCT06151132
Title: Treatment of Atrial Fibrillation in the Community Settings
Status: Completed | Type: Observational
Sponsor: ITMO University (Other)
Responsible Party: Principal Investigator, Artemiy Okhotin, researcher in Digital Public Health Technologies, ITMO University
Other Study IDs: ITMOU
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Atrial Arrhythmia; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Electric Countershock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with atrial fibrillation: Direct current cardioversion
  Interventions: Procedure: Direct current cardioversion

INTERVENTIONS:
Procedure: Direct current cardioversion — Direct current cardioversion to maintain sinus rhythm during rhythm control strategy

SUMMARY:
Description of treatment of cardiovascular diseases in community settings in Russia

DETAILED DESCRIPTION:
The study will describe different treatment modalities used in management of cardiovascular diseases in community hospital in small town of Tarusa in Russia. This part of the study will focus on atrial fibrillation and its treatment.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing direct current cardioversion for atrial fibrillation or flutter

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People receiving treatment for atrial fibrillation in Tarusa hospital.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Restoration of sinus rhythm | 1 day
  Restoration of sinus rhythm during direct current cardioversion
Maintenance in rhythm control strategy | 7 years
  Maintenance in rhythm control strategy during treatment of atrial fibrillation

OTHER OUTCOMES:
Gender | During procedure
  Gender
Age | During procedure
  Age
Body mass index | During procedure
  weight in kilograms divided by the square of height in meters
Heart Failure | Before procedure
  Past history of chronic heart failure
Arterial hypertension | Before procedure
  Past history of arterial hypertension
Coronary heart disease | Before procedure
  Past history of coronary heart disease
Diabetes mellitus | Before procedure
  Past history of diabetes mellitus
Type of arrhythmia | During procedure
  Atrial fibrillation or atrial flutter
Duration of arrhythmia | Before procedure
  Duration of episode of arrhythmia before cardioversion
Settings | During procedure
  Whether procedure performed in inpatient or outpatient settings
TEE | Before procedure
  Whether transesophageal echocardiography was performed before procedure
First procedure | Before procedure
  Whether it is the first cardioversion in the patient
Echo LVEF | During procedure
  Left ventricular ejection fraction measured by echocardiography
Echo LAVI | During procedure
  Left atrium volume index measured by echocardiography

IPD SHARING:
Plan to Share IPD: Yes
Deposition of all anonymized data in public repository.
Supporting Information: Analytic Code
Time Frame: With the publication, for 5 years.
Access Criteria: Public domain.